CLINICAL TRIAL: NCT07180979
Title: Comparison of Pericapsular Nerve Group (PENG) Block Versus Lumbar Erector Spinae Plane Block (L-ESPB) Combined With Sacral ESPB (S-ESPB) for Analgesia in Total Hip Arthroplasty (THA): A Randomized Clinical Trial
Brief Title: PENG vs L-ESPB With S-ESPB for Analgesia in Total Hip Arthroplasty
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 03/2025
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-09

CONDITIONS: Hip Osteoarthritis; Hip Arthropathy; Hip Pain Chronic
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Ropivacaine; Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): All participants will receive standard spinal anesthesia for total hip arthroplasty and multimodal postoperative analgesia according to institutional protocol.
  Interventions: Drug: Ropivacaine 0.5% Injectable Solution
- PENG + LFCN (Active Comparator): Participants in this group will receive an ultrasound-guided pericapsular nerve group (PENG) block combined with a lateral femoral cutaneous nerve (LFCN) block using local anesthetic. To preserve blinding, sham procedures will be performed at the lumbar and sacral erector spinae plane block sites (needle insertion and injection of 1-2 mL normal saline). Standard spinal anesthesia for total hip arthroplasty and multimodal postoperative analgesia will be administered as per institutional protocol.
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution
- L-ESPB + S-ESPB (Active Comparator): Participants in this group will receive ultrasound-guided lumbar erector spinae plane block (L-ESPB) combined with sacral erector spinae plane block (S-ESPB) using local anesthetic. To preserve blinding, sham procedures will be performed at the pericapsular and lateral femoral cutaneous nerve block sites (needle insertion and injection of 1-2 mL normal saline). Standard spinal anesthesia for total hip arthroplasty and multimodal postoperative analgesia will be provided according to institutional protocol.
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution

INTERVENTIONS:
Drug: Ropivacaine 0.5% Injectable Solution — All patients will receive standard spinal anesthesia with 0.5% ropivacaine, 10-15 mg intrathecally for total hip arthroplasty.
  Other Names: Spinal Anesthesia
  Arms: Control group
Drug: Ropivacaine 0.2% Injectable Solution — Ultrasound-guided pericapsular nerve group (PENG) block and lateral femoral cutaneous nerve (LFCN) block, with sham lumbar and sacral ESPBs.
  PENG block: 20 mL of 0.2% ropivacaine. LFCN block: 5 mL of 0.2% ropivacaine. Sham lumbar ESPB: 1-2 mL preservative-free normal saline at lumbar ESPB site. Sham sacral ESPB: 1-2 mL preservative-free normal saline at sacral ESPB site. All patients will receive standard spinal anesthesia with 0.5% ropivacaine, 10-15 mg intrathecally for total hip arthroplasty.
  Arms: PENG + LFCN
Drug: Ropivacaine 0.2% Injectable Solution — Ultrasound-guided lumbar erector spinae plane block (L-ESPB) and sacral erector spinae plane block (S-ESPB), with sham PENG and LFCN blocks.
  Lumbar ESPB: 20 mL of 0.2% ropivacaine at L3 transverse process level. Sacral ESPB: 20 mL of 0.2% ropivacaine at sacral intermediate crest. Sham PENG block: 1-2 mL preservative-free normal saline at PENG site. Sham LFCN block: 1-2 mL preservative-free normal saline at LFCN site. All patients will receive standard spinal anesthesia with 0.5% ropivacaine, 10-15 mg intrathecally for total hip arthroplasty.
  Arms: L-ESPB + S-ESPB

SUMMARY:
The goal of this clinical trial is to evaluate whether different types of regional anesthesia can improve pain control and functional recovery after total hip arthroplasty in adult patients undergoing elective hip replacement surgery.

The main questions it aims to answer are:

Does the PENG block reduce opioid use in the first 48 hours after surgery more effectively than the combined L-ESPB + S-ESPB technique? Which method provides better pain relief, preserves muscle strength, and supports earlier mobilization? Researchers will compare the Pericapsular Nerve Group (PENG) block with the combination of Lumbar and Sacral Erector Spinae Plane Blocks (L-ESPB + S-ESPB) to see which provides better pain control, fewer side effects, and faster recovery.

Participants will:

Be randomly assigned to receive one of the two types of ultrasound-guided regional anesthesia Undergo standard hip replacement surgery under spinal anesthesia Be monitored for pain scores, opioid use, time to first walking, muscle strength, satisfaction, and side effects over the first 48 hours after surgery.

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) is associated with moderate-to-severe postoperative pain, which can impair early mobilization and functional recovery. Regional anesthesia techniques, such as the pericapsular nerve group (PENG) block and the erector spinae plane (ESP) block, have been introduced as motor-sparing alternatives to femoral and lumbar plexus blocks. The PENG block targets articular branches of the femoral, obturator, and accessory obturator nerves, offering effective analgesia with minimal motor blockade. Meanwhile, the lumbar ESPB (L-ESPB) and sacral ESPB (S-ESPB) may provide a broader, yet still motor-sparing, analgesic field by targeting both lumbar and sacral nerve roots involved in hip innervation.

To date, no randomized trial has compared PENG with a dual-level ESP block approach (L-ESPB + S-ESPB) in THA patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* ASA physical status I-III
* Elective unilateral THA via posterior or lateral approach
* Informed consent provided

Exclusion Criteria:

* Allergy to study drugs (ropivacaine, dexamethasone)
* Chronic opioid use (>30 MME/day)
* Coagulopathy or infection at the injection site
* BMI > 40 kg/m²
* Pre-existing motor weakness or neuropathy in the affected limb
* Cognitive impairment precluding informed consent

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Total opioid consumption | first 48 hours postoperatively
  morphine milligram equivalents (MME)

SECONDARY OUTCOMES:
Pain scores | 4 hours after surgery
  Numeric Rating Scale (NRS), ranging from 0 ("no pain") to 10 ("the worst pain imaginable")- at rest and during mobilization
Pain scores | 8 hours after surgery
  Numeric Rating Scale (NRS), ranging from 0 ("no pain") to 10 ("the worst pain imaginable")- at rest and during mobilization
Pain scores | 12 hours after surgery
  Numeric Rating Scale (NRS), ranging from 0 ("no pain") to 10 ("the worst pain imaginable")- at rest and during mobilization
Pain scores | 24 hours after surgery
  Numeric Rating Scale (NRS), ranging from 0 ("no pain") to 10 ("the worst pain imaginable")- at rest and during mobilization
Pain scores | 48 hours after surgery
  Numeric Rating Scale (NRS), ranging from 0 ("no pain") to 10 ("the worst pain imaginable")- at rest and during mobilization
Time to ambulation | 48 hours after surgery
  Time to ambulation is defined as the time interval (in hours) from the end of surgery (skin closure) to the patient's first successful attempt at ambulation with or without assistance, as determined by the attending physiotherapist or nursing staff.
Quadriceps muscle strength | 4 hours after surgery
  Quadriceps muscle strength assessed using medical research council scale [range 0:5]
Quadriceps muscle strength | 8 hours after surgery
  Quadriceps muscle strength assessed using medical research council scale [range 0:5]
Quadriceps muscle strength | 12 hours after surgery
  Quadriceps muscle strength assessed using medical research council scale [range 0:5]
Quadriceps muscle strength | 24 hours after surgery
  Quadriceps muscle strength assessed using medical research council scale [range 0:5]
Quadriceps muscle strength | 48 hours after surgery
  Quadriceps muscle strength assessed using medical research council scale [range 0:5]

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Reysner, Study Chair — Poznan University of Medical Sciences; Tomasz Reysenr, M.D., Principal Investigator — Poznan Univesity of Medical Sciences

IPD SHARING:
Plan to Share IPD: Yes